CLINICAL TRIAL: NCT01507506
Title: Phase III Randomized Study Comparing 2 Brain Conformational Radiotherapy in Combination With Chemotherapy in the Treatment of Glioblastoma : Standard 3D Conformational Radiotherapy Versus Intensity-modulated Radiotherapy With Simultaneous-integrated Boost Guided by Magnetic Resonance Spectroscopic Imaging
Brief Title: Phase III Study Comparing 2 Brain Conformational Radiotherapy in Combination With Chemotherapy in the Treatment of Glioblastoma
Acronym: SPECTRO GLIO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08 TETE 01
Record Dates: First submitted 2011-12-20; First posted 2012-01-11 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Radiotherapy; Intensity modulated radiation therapy (IMRT); Magnetic resonance spectroscopic imaging (MRSI)
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional arm (Active Comparator): 3-dimensional conformal radiotherapy + Temozolomide
  Interventions: Radiation: Radiotherapy
- Experimental arm (Experimental): simultaneous-integrated boost with intensity-modulated radiotherapy guided by magnetic resonance spectroscopic imaging + Temozolomide
  Interventions: Radiation: Experimental arm

INTERVENTIONS:
Radiation: Radiotherapy — Conventional arm: 3D conformational radiotherapy (arm A): 60 Gy per fractions of 2 Gy in 30 sessions on the PTV1 (contrast enhancement + 2 cm) with a linear accelerator equipped with a portal imaging.
  +
  Chemotherapy (Drug) :treatment should be combined with temozolomide during and after radiotherapy in a conventional treatment Stupp (Stupp et al. 2005), ie :
  * during radiotherapy : Temozolomide 75 mg/m2/day by oral route every day,
  * post radiotherapy : 6 cycles of Temozolomide oral route : 150 mg/m2/day from D1 to D5 for the 1st cycle followed by 200 mg/m2/day from D28 to D32.
  Arms: Conventional arm
Radiation: Experimental arm — Conformational radiotherapy with simultaneous integrated boost by intensity modulation (Arm B): 60 Gy per fraction of 2 Gy in 30 sessions on the PTV1 (contrast enhancement + 2 cm) with concomitant daily superimposed boost on spectroscopic active region (PTV2) corresponding to the ratio Cho / NAA> 2 + 0.7 mm + contrast enhancement + 3mm. The PTV2 will receive a daily dose of 2.4 Gy for a cumulative dose of 72 Gy Only irradiation with simultaneous integrated boost are allowed
  +
  Chemotherapy (Drug) :treatment should be combined with temozolomide during and after radiotherapy in a conventional treatment Stupp (Stupp et al. 2005), ie :
  * during radiotherapy : Temozolomide 75 mg/m2/day by oral route every day,
  * post radiotherapy : 6 cycles of Temozolomide oral route : 150 mg/m2/day from D1 to D5 for the 1st cycle followed by 200 mg/m2/day from D28 to D32.
  Arms: Experimental arm

SUMMARY:
This is a multi-institutional phase III clinical study of interventional type. The trial will include 220 patients with confirmed unifocal glioblastoma over a period of 3 years + 3 years of follow up.

Patients with unifocal glioblastoma (diagnosis confirmed by histology on tumoral biopsy or surgical specimen) and who meet all eligibility criteria will be randomized in one chemoradiotherapy arm :

* Conventional arm: 3-dimensional conformational radiotherapy + Temozolomide
* Experimental arm : simultaneous-integrated boost with intensity-modulated radiotherapy guided by magnetic resonance spectroscopic imaging + Temozolomide The patient monitoring will be regular and standardized. The main objective of this study is to improve overall survival of patients treated in experimental group (with simultaneous integrated boost).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have unifocal glioblastoma (grade IV astrocytoma, WHO classification). The GBM can be:

   * Or resectable and the patient has received curative surgery
   * Or unresectable, and the largest tumor diameter (contrast enhancement) must be less than 5 cm on MRI
2. In all cases, the diagnosis must be confirmed by a pathologist. In patients for whom surgery is not possible, the diagnosis is confirmed by a biopsy of tumor tissue.
3. Methylation status of MGMT gene promoter is known
4. Patients who have undergone resection should have received an MRI or a scan after surgery in order to visualize residual tumor. If not, the operative report must be available.
5. Surgery or biopsy must have occurred 45 days before the start of radiotherapy.
6. WHO ≤ 2
7. Age ≥ 18 years
8. Signed Consent collected before any specific procedure in the study
9. Patient member in a national insurance scheme

Exclusion Criteria:

1. Signs of hemorrhage on pre-radiotherapy MRI preventing a good spectrometric analysis
2. Patient with multifocal glioblastoma
3. Tumor located within 2 cm of the optic chiasm
4. Patient with leptomeningeal metastases,
5. patients prone to epileptic seizures despite treatment with anticonvulsant
6. Patients who received other previous treatment for glioblastoma multiforme
7. Abnormal haematological results at inclusion with:

   * Neutrophils < 1500/mm3
   * Blood-platelets < 100000/mm3
8. Severe or chronic renal insufficiency (creatinin clearance ≤ 30 ml/min calculated using Cockroft-Gault's formula
9. Patient unable to follow procedures, visits, examinations described in the study
10. Any usual formal indication against imaging examinations (important claustrophobia, pace maker ...)
11. Pregnant women or nursing mothers can not participate in the study. Women of childbearing age must have a negative pregnancy test within 72 hours prior to study entry
12. Men and women of childbearing age must use effective contraception at study entry and throughout the study
13. Any concomitant or previous malignant disease within 5 years prior to study entry
14. Any prior systemic chemotherapy within 5 years prior to inclusion (for malignant disease in medical history)
15. Any other medical conditions making the inclusion of the patient in the study inappropriate in the opinion of the investigator
16. Patient under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Overall survival defined as the time from randomization to the date of death or date of last follow-up news (censured data) | 8 years

SECONDARY OUTCOMES:
Progression-free survival, defined as the time from randomization to the date of progression or death | 8 years
Safety evaluated according to the classification of NCI CTCAE (Common Terminology Criteria for Adverse Events)V3.0 | 8 years

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Clinique Claude Bernard, Albi
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Hospices Civils de Lyon (Hôpital Lyon Sud/Hôpital P. Wertheimer), Lyon
  - Centre Leon Berard, Lyon
  - AP HM - Hôpital La Timone, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Institut de Cancerologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - CHU de Strasbourg, Strasbourg
  - Institut Claudius REGAUD, Toulouse
  - Centre Marie Curie, Valence

REFERENCES:
- [Derived] Laprie A, Noel G, Chaltiel L, Truc G, Sunyach MP, Charissoux M, Magne N, Auberdiac P, Biau J, Ken S, Tensaouti F, Khalifa J, Sidibe I, Roux FE, Vieillevigne L, Catalaa I, Boetto S, Uro-Coste E, Supiot S, Bernier V, Filleron T, Mounier M, Poublanc M, Olivier P, Delord JP, Cohen-Jonathan-Moyal E. Randomized phase III trial of metabolic imaging-guided dose escalation of radio-chemotherapy in patients with newly diagnosed glioblastoma (SPECTRO GLIO trial). Neuro Oncol. 2024 Jan 5;26(1):153-163. doi: 10.1093/neuonc/noad119. PMID 37417948
- [Derived] Laprie A, Ken S, Filleron T, Lubrano V, Vieillevigne L, Tensaouti F, Catalaa I, Boetto S, Khalifa J, Attal J, Peyraga G, Gomez-Roca C, Uro-Coste E, Noel G, Truc G, Sunyach MP, Magne N, Charissoux M, Supiot S, Bernier V, Mounier M, Poublanc M, Fabre A, Delord JP, Cohen-Jonathan Moyal E. Dose-painting multicenter phase III trial in newly diagnosed glioblastoma: the SPECTRO-GLIO trial comparing arm A standard radiochemotherapy to arm B radiochemotherapy with simultaneous integrated boost guided by MR spectroscopic imaging. BMC Cancer. 2019 Feb 21;19(1):167. doi: 10.1186/s12885-019-5317-x. PMID 30791889
- [Derived] Ken S, Deviers A, Filleron T, Catalaa I, Lotterie JA, Khalifa J, Lubrano V, Berry I, Peran P, Celsis P, Moyal EC, Laprie A. Voxel-based evidence of perfusion normalization in glioblastoma patients included in a phase I-II trial of radiotherapy/tipifarnib combination. J Neurooncol. 2015 Sep;124(3):465-73. doi: 10.1007/s11060-015-1860-8. Epub 2015 Jul 19. PMID 26189058